CLINICAL TRIAL: NCT02669953
Title: Response to Aflibercept After Previous Intravitreal Ranibizumab Treatment in Neovascular Age-Related Macular Degeneration
Brief Title: Aflibercept in Recurrent or Persistent CNV
Acronym: OPHTH-010915
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Prof. PD. Dr., Medical University of Vienna
Other Study IDs: OPHTH-010915 (Ex-Oct)
Record Dates: First submitted 2016-01-18; First posted 2016-02-01 (Estimated); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Age Related Macular Degeneration; Intravitreal Injections; Diabetic Macular Edema
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- AMD patients previously teated with Lucentis: Adults ≥ 50 years; Patients who have been treated with ranibizumab due to wet age-related macular degeneration for up to one year; Patients who have a BCVA score better than 20/400 in the study eye using ETDRS; Willingness and ability to comply with regular visits; Signed informed consent form;
  The patient can take his medicine in the prescribed manner. The prescribed drugs do not constitute an exclusion criteria.
  Interventions: Drug: Aflibercept
- treatment naive AMD patients: Adults ≥ 50 years; Patients who have a BCVA score better than 20/400 in the study eye using ETDRS;
  Interventions: Drug: Aflibercept
- DME patients previously teated with Lucentis: Adults ≥ 50 years; Patients who have been treated with ranibizumab due to DME for up to one year; Patients who have a BCVA score better than 20/400 in the study eye using ETDRS;
  Interventions: Drug: Aflibercept
- treatment naive DME patients: Adults ≥ 50 years; Patients who have a BCVA score better than 20/400 in the study eye using ETDRS;
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept

SUMMARY:
Age-related macular degeneration (AMD) and diabetic retinopathy are among the most common disorders causing visual disability in elderly people. AMD leads to dysfunction and loss of photoreceptors in the central retina. Neovascular AMD (nAMD) affects visual function early in the disease process.

The purpose of the study is to evaluate the effect of switching from ranibizumab therapy to the current routine therapy using aflibercept in eyes with treatment naive, recurrent or persistent nAMD, treatment naive diabetic retinopathy and pretreated diabetic retinopathy.

20 patients with recurrent or persistent nAMD, previously treated with intravitreal ranibizumab for up to one year will be included in this trial. Patients will be examined in monthly intervals over 12 months follow-up.

Examinations carried out will include: Best-corrected visual acuity (BCVA) using ETDRS charts at 4m distance, Reading Performance (RP), Standard ophthalmic examinations (SOE incl. funduscopy and applanation tonometry), Optical coherence tomography (OCT), Autofluorescence fundus image (AF) & red-free autofluorescence fundus image (RF), Color fundus photography (CFP), Fluorescein angiography and indocyaningreen angiography (FLA/ICG), Microperimetry (MP), as well as Non-invasive OCT based optical angiography (AngioVue).

ELIGIBILITY:
Inclusion Criteria:

Adults ≥ 50 years

* Patients who have been treated with ranibizumab due to wet age-related macular degeneration for up to one year
* BCVA >= 20/400 in the study eye using ETDRS
* Willingness and ability to comply with regular visits
* Signed informed consent

Exclusion Criteria:

* Any surgical treatment of the eye within 3 months prior to baseline in the study eye
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma mediation)
* Aphakia or absence of the posterior capsule (excluding YAG-capsulotomy) in the study eye
* Retinal pigment epithelial tear involving the macula in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 Patients with nAMD
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent change in Best-Corrected Visual Acuity (BCVA) | After one year compared to baseline
Anatomic changes in the macula as assessed with OCT (central retinal thickness, morphologic changes, fundus photos) | after one year compared to baseline

SECONDARY OUTCOMES:
Number of retreatments | after one year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No